CLINICAL TRIAL: NCT01421342
Title: CSP #576 - VA Augmentation and Switching Treatments for Improving Depression Outcomes (VAST-D)
Brief Title: VA Augmentation and Switching Treatments for Improving Depression Outcomes
Acronym: VAST-D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 576
Record Dates: First submitted 2011-08-05; First posted 2011-08-22 (Estimated); Results first posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-04

CONDITIONS: Major Depressive Disorder
Keywords: Mood Disorder; Depression; Depressive Disorder; Depressive Disorder, Major; Bupropion; Aripiprazole; Remission; Relapse; Cost-Effectiveness; Atypical Antipsychotic; Antidepressant; Augmentation; Veterans; Mental Health
MeSH Terms: conditions — Depressive Disorder, Major; Mood Disorders; Depression; Depressive Disorder; Recurrence; Psychological Well-Being | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Switching: Bupropion-SR (Active Comparator): Switching: Bupropion-SR
  Interventions: Drug: Switching: Bupropion-SR
- Augmenting: Antidepressant + Bupropion-SR (Active Comparator): Augmenting: Antidepressant + Bupropion-SR
  Interventions: Drug: Augmenting: Antidepressant + Bupropion-SR
- Augmenting: Antidepressant + Aripiprazole (Active Comparator): Augmenting: Antidepressant + Aripiprazole
  Interventions: Drug: Augmenting: Antidepressant + Aripiprazole

INTERVENTIONS:
Drug: Switching: Bupropion-SR — Bupropion-SR (Dose: 150 mg - 400 mg taken per day orally for up to 36 weeks): Initiating with bupropion-SR dose of 150 mg, then increasing dose per protocol up to 400 mg (200 mg BID), maintaining or decreasing dose for up to 36 weeks depending on response and side effect profile through the acute and continuation phases.
  Arms: Switching: Bupropion-SR
Drug: Augmenting: Antidepressant + Bupropion-SR — Current antidepressant (either a SSRI or a SNRI or mirtazapine): Continue the dose prescribed at time of enrollment, or adjust depending on response or side effect profile for up to 36 weeks.
  And
  Bupropion-SR (Dose: 150 mg - 400 mg taken per day orally for up to 36 weeks): Initiating with bupropion-SR dose of 150 mg, then increasing dose per protocol up to 400 mg (200 mg BID), maintaining or decreasing dose for up to 36 weeks depending on response and side effect profile through the acute and continuation phases.
  Arms: Augmenting: Antidepressant + Bupropion-SR
Drug: Augmenting: Antidepressant + Aripiprazole — Current antidepressant (either a SSRI or a SNRI or mirtazapine): Continue the dose prescribed at time of enrollment or adjust depending on response or side effect profile for up to 36 weeks.
  And
  Aripiprazole (Dose: 2 mg - 15 mg taken orally once per day for up to 36 weeks): Initiating with aripiprazole dose of 2 mg for one week, then increasing dose per protocol up to 15 mg, maintaining or decreasing dose for up to 36 weeks depending on response and side effect profile through the acute and continuation phases.
  Arms: Augmenting: Antidepressant + Aripiprazole

SUMMARY:
The overall purpose is to determine research based 'next-steps' for outpatients with major depressive disorder who have not had satisfactory outcomes to standard 'first-step' treatments. The primary objective is to compare the acute (up to 12 weeks) treatment effectiveness of augmenting an antidepressant with aripiprazole or with bupropion-slow release (SR) vs. switching treatment to bupropion-SR monotherapy on symptom remission in Veterans with Major Depressive Disorder (MDD) who have not achieved optimal response after an adequate trial on antidepressant (a selective serotonin reuptake inhibitor [SSRI] or serotonin and norepinephrine reuptake inhibitor [SNRI] or mirtazapine) monotherapy. The secondary objectives are to compare the acute (up to 12 weeks) and long term (up to 36 weeks) efficacy, safety, effects on functioning, suicidality, quality of life, anxiety and other associated symptoms, costs and cost-effectiveness of each of the three treatments.

DETAILED DESCRIPTION:
The overall aim of VAST-D is to enhance treatment outcomes for representative outpatients diagnosed with nonpsychotic major depressive disorder (MDD) and treated in primary or psychiatric VA care settings. In particular, VAST-D is designed to determine the comparative effectiveness of different treatment options for participants with MDD who fail to have a satisfactory outcome to treatment with their initial antidepressants.

These options may be conceptualized as representing two overall treatment strategies: 1) Medication Switch - switching from the initial antidepressant to another antidepressant medication, specifically bupropion-SR and 2) Medication Augmentation - augmenting the initial antidepressant with a second antidepressant, specifically bupropion-SR or a second generation antipsychotic, specifically aripiprazole. VAST-D's primary goal is to determine which of these 3 treatment strategies is most likely to lead to remission. Other key objectives include comparisons of response, time to remission, time to response, relapse, anxiety symptoms, suicidal ideation and behaviors, side effects, tolerability, quality of life, health related costs and satisfaction with participation in the study.

VAST-D will enroll 1518 total patients of both genders and all ethnic/racial and socioeconomic backgrounds. All patients will meet Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV-TR (text revised) criteria for nonpsychotic MDD. The diagnostic criteria for eligibility will be established by clinical interview supplemented with the 9-item Patient Health Questionnaire (PHQ-9). Final determination for eligibility will be made by the study clinician. Only participants with a suboptimal outcome to a well documented, adequately delivered (dose and duration), trial with selective serotonin reuptake inhibitor (SSRI) or a serotonin and norepinephrine reuptake inhibitor (SNRI) or mirtazapine will be eligible for the study. Failure to achieve an adequate outcome will be ascertained by a score on the 16-item Quick Inventory of Depressive Symptomatology - Clinician rated (QIDS-C16) scale >= 16 (considered severe depression) after at least 6 weeks of treatment or QIDS-C16 >= 11 (considered moderately severe depression) after at least 8 weeks of treatment. Otherwise, the inclusion criteria are broad and the exclusion criteria are few; participants with most comorbid general medical or psychiatric disorders are generally included to provide a broadly representative sample.

Participants will be randomized (1:1:1 ratio) to switch to bupropion-SR alone (n=506), current antidepressant plus bupropion-SR (n=506), or current antidepressant plus aripiprazole (n=506). Treatment will be guided by clinician-rated symptom measures (the PHQ-9) and global side effects measures (the Frequency, Intensity, and Burden of Side Effects Rating or FIBSER) obtained at each treatment visit. Acute treatment visits will occur at baseline and at weeks 1, 2, 4, 6, 8, 10, and 12 to ensure delivery of appropriate and yet vigorous and tolerable pharmacotherapy. Participants who tolerate the acute treatment and achieve adequate response at 12 weeks will enter the 24-week Continuation Treatment phase, during which the initial treatment will continue and visits will occur every four weeks subsequently until patients have been followed for 36 weeks post-randomization. The QIDS-C16 will be administered at baseline and at each follow-up visit by an independent evaluator (who will be blinded to treatment assignment) to measure symptoms of depression for the study outcomes of remission, response and relapse. Neither the participant nor the treating clinician will be blinded to treatment.

Primary hypotheses:

Primary hypothesis 1.a: Remission rate from major depressive disorder will be higher in patients whose treatment is augmented with bupropion-SR (antidepressant + bupropion-SR) compared to those switched to bupropion-SR monotherapy.

Primary Hypothesis 1.b: Remission rate from major depressive disorder will be higher in patients whose treatment is augmented with aripiprazole (antidepressant + aripiprazole) compared to those switched to bupropion-SR monotherapy.

Secondary hypotheses:

Secondary Hypothesis 2.a: Remission rate will be greater in patients whose treatment is augmented with bupropion-SR (antidepressant + bupropion-SR) than in those augmented with aripiprazole (antidepressant + aripiprazole).

Secondary Hypothesis 2.b: Relapse rate (within 36 weeks of the initiation of treatment) will be lower in patients whose antidepressant is augmented with bupropion-SR (antidepressant + bupropion-SR) than in those whose antidepressant is switched to bupropion-SR monotherapy.

Secondary Hypothesis 2.c: Relapse rate (within 36 weeks of the initiation of treatment) will be lower in patients whose treatment is augmented with aripiprazole (antidepressant + aripiprazole) vs. those switched to bupropion-SR monotherapy.

Secondary Hypothesis 2.d: Relapse rate (within 36 weeks of the initiation of treatment) will be lower in patients whose treatment is augmented with bupropion-SR (antidepressant + bupropion-SR) than in patients whose treatment was augmented with aripiprazole (antidepressant + aripiprazole).

Secondary Hypothesis 2.e: The proportion of patients who develop akathisia, other akathisia-like side effects (e.g., tremor, irritability, motor restlessness) and extrapyramidal side effects will be greater in the patients whose antidepressant treatment is augmented with aripiprazole (antidepressant + aripiprazole) compared to patients whose treatment is augmented with bupropion-SR (antidepressant + bupropion-SR), or switched to bupropion-SR monotherapy.

Secondary Hypothesis 2.f: The relative costs (direct and indirect) of augmenting an antidepressant with aripiprazole (antidepressant + aripiprazole) will be greater than the costs of antidepressant augmentation with bupropion-SR (antidepressant + bupropion-SR), and the costs of antidepressant augmentation with bupropion-SR (antidepressant + bupropion-SR) will be greater than the costs of switching to bupropion-SR monotherapy, and augmentation and monotherapy with bupropion-SR will be more cost-effective than aripiprazole augmentation.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of single or recurrent, non-psychotic, major depressive disorder
* Currently taking a selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) or mirtazapine for major depressive disorder
* Need for "next-step" treatment based on documented suboptimal outcome from current antidepressant treatment for major depressive episode (at least 6 weeks treatment with a QIDS-C16 >= 16 or at least 8 weeks with a QIDS-C16 >= 11; and at least 3 weeks at a stable "optimal" dose
* Age: 18 years of age or older

Exclusion Criteria:

* Prior inadequate response after an adequate treatment trial or clear cut intolerance to either of the study medications (aripiprazole or bupropion)
* Current treatment with bupropion, aripiprazole or any other antipsychotic agent
* Lifetime history of bipolar disorder, schizophrenia, schizoaffective disorder, or psychosis not otherwise specified
* Current diagnosis of Dementia
* Current diagnosis of an eating disorder or a seizure disorder
* High suicide risk currently requiring acute intervention (other than outpatient treatment of depression)
* Unstable, serious medical condition or one requiring acute medical treatment, or anticipation of hospitalization for extended care
* Requiring immediate hospitalization for psychiatric disorders
* Physiologic substance dependence requiring detoxification (excluding nicotine) in the past 30 days (substance abuse is not an exclusion criteria)
* Taking any concomitant medication that contraindicates any of treatment options or augmenting agents known to have an antidepressant effect
* Concurrent or recent participation (within the last 30 days) in another conflicting clinical trial with a mental health, investigational drug, or medical device intervention
* Female - pregnant or lactating or planning to become pregnant
* Patient was not able or willing to provide informed consent; or changed mind about participating prior to randomization
* Patient was not referred to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1522 (Actual)
Dates: Start 2012-12; Primary Completion 2015-08 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Somaia Mohamed, PhD, Study Chair — VA Connecticut Healthcare System West Haven Campus, West Haven, CT; Sidney Zisook, MD, Study Chair — VA San Diego Healthcare System, San Diego, CA
Locations (35):
- United States (35):
  - Tuscaloosa VA Medical Center, Tuscaloosa, AL, Tuscaloosa, Alabama
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tucson, Tucson, Arizona
  - VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Kansas City VA Medical Center, Kansas City, MO, Kansas City, Missouri
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri
  - Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico
  - Asheville VA Medical Center, Asheville, NC, Asheville, North Carolina
  - Salisbury W.G. (Bill) Hefner VA Medical Center, Salisbury, NC, Salisbury, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Philadelphia VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Memphis VA Medical Center, Memphis, TN, Memphis, Tennessee
  - Central Texas Veterans Health Care System, Temple, TX, Temple, Texas
  - Salem VA Medical Center, Salem, VA, Salem, Virginia
  - VA Puget Sound Health Care System American Lake Division, Tacoma, WA, Tacoma, Washington
  - Clarksburg Louis A. Johnson VA Medical Center, Clarksburg, WV, Clarksburg, West Virginia
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin
  - Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohamed S, Johnson GR, Vertrees JE, Guarino PD, Weingart K, Young IT, Yoon J, Gleason TC, Kirkwood KA, Kilbourne AM, Gerrity M, Marder S, Biswas K, Hicks P, Davis LL, Chen P, Kelada A, Huang GD, Lawrence DD, LeGwin M, Zisook S. The VA augmentation and switching treatments for improving depression outcomes (VAST-D) study: Rationale and design considerations. Psychiatry Res. 2015 Oct 30;229(3):760-70. doi: 10.1016/j.psychres.2015.08.005. Epub 2015 Aug 6. PMID 26279130
- [Result] Zisook S, Tal I, Weingart K, Hicks P, Davis LL, Chen P, Yoon J, Johnson GR, Vertrees JE, Rao S, Pilkinton PD, Wilcox JA, Sapra M, Iranmanesh A, Huang GD, Mohamed S. Characteristics of U.S. Veteran Patients with Major Depressive Disorder who require "next-step" treatments: A VAST-D report. J Affect Disord. 2016 Dec;206:232-240. doi: 10.1016/j.jad.2016.07.023. Epub 2016 Jul 26. PMID 27479536
- [Result] Mohamed S, Johnson GR, Chen P, Hicks PB, Davis LL, Yoon J, Gleason TC, Vertrees JE, Weingart K, Tal I, Scrymgeour A, Lawrence DD, Planeta B, Thase ME, Huang GD, Zisook S; and the VAST-D Investigators; Rao SD, Pilkinton PD, Wilcox JA, Iranmanesh A, Sapra M, Jurjus G, Michalets JP, Aslam M, Beresford T, Anderson KD, Fernando R, Ramaswamy S, Kasckow J, Westermeyer J, Yoon G, D'Souza DC, Larson G, Anderson WG, Klatt M, Fareed A, Thompson SI, Carrera CJ, Williams SS, Juergens TM, Albers LJ, Nasdahl CS, Villarreal G, Winston JL, Nogues CA, Connolly KR, Tapp A, Jones KA, Khatkhate G, Marri S, Suppes T, LaMotte J, Hurley R, Mayeda AR, Niculescu AB 3rd, Fischer BA, Loreck DJ, Rosenlicht N, Lieske S, Finkel MS, Little JT. Effect of Antidepressant Switching vs Augmentation on Remission Among Patients With Major Depressive Disorder Unresponsive to Antidepressant Treatment: The VAST-D Randomized Clinical Trial. JAMA. 2017 Jul 11;318(2):132-145. doi: 10.1001/jama.2017.8036. PMID 28697253
- [Derived] Zisook S, Johnson GR, Planeta B, Mohamed S. How Does Positive Mental Health Affect Next-Step Treatment Outcomes in Treatment-Resistant Depression? A VAST-D Report. J Clin Psychopharmacol. 2025 Sep-Oct 01;45(5):421-431. doi: 10.1097/JCP.0000000000002051. Epub 2025 Jul 31. PMID 40742171
- [Derived] Zisook S, Planeta B, Hicks PB, Chen P, Davis LL, Villarreal G, Sapra M, Johnson GR, Mohamed S. Childhood adversity and adulthood major depressive disorder. Gen Hosp Psychiatry. 2022 May-Jun;76:36-44. doi: 10.1016/j.genhosppsych.2022.03.008. Epub 2022 Mar 24. PMID 35366613
- [Derived] Zisook S, Johnson GR, Hicks P, Chen P, Beresford T, Michalets JP, Rao S, Thase ME, Wilcox J, Sevilimedu V, Mohamed S. Continuation phase treatment outcomes for switching, combining, or augmenting strategies for treatment-resistant major depressive disorder: A VAST-D report. Depress Anxiety. 2021 Feb;38(2):185-195. doi: 10.1002/da.23114. Epub 2020 Nov 22. PMID 33225492
- [Derived] Mohamed S, Johnson GR, Sevilimedu V, Rao SD, Hicks PB, Chen P, Lauro K, Jurjus G, Pilkinton P, Davis L, Wilcox JA, Iranmanesh A, Sapra M, Aslam M, Michalets J, Thase M, Zisook S; CSP#576 VAST-D Investigators. Impact of Concurrent Posttraumatic Stress Disorder on Outcomes of Antipsychotic Augmentation for Major Depressive Disorder With a Prior Failed Treatment: VAST-D Randomized Clinical Trial. J Clin Psychiatry. 2020 Jun 23;81(4):19m13038. doi: 10.4088/JCP.19m13038. PMID 32603560
- [Derived] Zisook S, Johnson GR, Tal I, Hicks P, Chen P, Davis L, Thase M, Zhao Y, Vertrees J, Mohamed S. General Predictors and Moderators of Depression Remission: A VAST-D Report. Am J Psychiatry. 2019 May 1;176(5):348-357. doi: 10.1176/appi.ajp.2018.18091079. Epub 2019 Apr 5. PMID 30947531
- [Derived] Yoon J, Zisook S, Park A, Johnson GR, Scrymgeour A, Mohamed S. Comparing Cost-Effectiveness of Aripiprazole Augmentation With Other "Next-Step" Depression Treatment Strategies: A Randomized Clinical Trial. J Clin Psychiatry. 2018 Dec 18;80(1):18m12294. doi: 10.4088/JCP.18m12294. PMID 30695291

RESULTS

PARTICIPANT FLOW:
Period: Acute Treatment Phase (12 Weeks)
Arm/Group | Switching: Bupropion-SR | Augmenting: Antidepressant + Bupropion-SR | Augmenting: Antidepressant + Aripiprazole
Started | 511 | 506 | 505
Completed | 353 | 378 | 406
Not Completed | 158 | 128 | 99
Not completed — Lack of Efficacy | 49 | 28 | 13
Not completed — Adverse Event | 53 | 38 | 27
Not completed — Withdrawal by Subject | 23 | 20 | 13
Not completed — Death | 0 | 0 | 3
Not completed — Lost to Follow-up | 6 | 18 | 21
Not completed — Non-adherence | 15 | 7 | 13
Not completed — Dure to other illness | 3 | 2 | 4
Not completed — Participant moved away | 1 | 6 | 1
Not completed — Other reason for withdrawal | 8 | 9 | 4
Period: Completed to Week 12 But Then Withdrawn
Arm/Group | Switching: Bupropion-SR | Augmenting: Antidepressant + Bupropion-SR | Augmenting: Antidepressant + Aripiprazole
Started | 353 | 378 | 406
Completed | 204 | 253 | 268
Not Completed | 149 | 125 | 138
Not completed — Lack of Efficacy | 111 | 93 | 88
Not completed — QIDS Score >=11 | 7 | 10 | 12
Not completed — Adverse Event | 4 | 3 | 6
Not completed — Withdrawal by Subject | 13 | 4 | 11
Not completed — Lost to Follow-up | 4 | 3 | 3
Not completed — Non-adherence | 5 | 4 | 5
Not completed — Due to Other Illness | 1 | 0 | 2
Not completed — Participant Moved Away | 1 | 5 | 5
Not completed — Oher reason for withdrawal | 3 | 3 | 4
Not completed — End of Study Time | 0 | 0 | 2
Period: Continuation of Treatment (Week 12 - 36)
Arm/Group | Switching: Bupropion-SR | Augmenting: Antidepressant + Bupropion-SR | Augmenting: Antidepressant + Aripiprazole
Started | 204 | 253 | 268
Completed | 152 | 194 | 203
Not Completed | 52 | 59 | 65
Not completed — Lack of Efficacy | 11 | 5 | 11
Not completed — Adverse Event | 0 | 6 | 11
Not completed — Withdrawal by Subject | 7 | 6 | 4
Not completed — Lost to Follow-up | 4 | 11 | 9
Not completed — Non-adherence | 3 | 8 | 4
Not completed — End of Study Time | 15 | 20 | 14
Not completed — Participant moved away | 4 | 1 | 3
Not completed — Due to Other Illness | 2 | 2 | 2
Not completed — Other reason for withdrawal | 6 | 0 | 7

BASELINE CHARACTERISTICS:
Population: The ASEX (female) version of the questionnaire was specific to females.The ASEX (male) version of the questionnaire was specific to males. Not all females or males completed the questionnaire, therefore, the number of responders is lower than number of participants due to missing responses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Switching: Bupropion-SR | Augmenting: Antidepressant + Bupropion-SR | Augmenting: Antidepressant + Aripiprazole | Total
Number analyzed (Participants) | 511 | 506 | 505 | 1522
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (12.2) | 54.4 (12.2) | 54.2 (12.3) | 54.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 81 | 77 | 226
  Male | 443 | 425 | 428 | 1296
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 3
  Not Hispanic or Latino | 454 | 449 | 459 | 1362
  Unknown or Not Reported | 57 | 55 | 45 | 157
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 8 | 6 | 22
  Asian | 2 | 1 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 1 | 5
  Black or African American | 129 | 115 | 126 | 370
  White | 341 | 343 | 338 | 1022
  More than one race | 10 | 20 | 13 | 43
  Unknown or Not Reported | 19 | 17 | 17 | 53
QIDS-C16 Score [Mean (Standard Deviation); unit: units on a scale] — Quick Inventory of Depression Symptomatology - Clinician rated (QIDS-C16) score: summary score of severity of depression symptoms. (range: 0 [better],27 [worse]), www.ids-qids.org
  units on a scale | 16.6 (3.3) | 16.6 (3.2) | 16.9 (3.3) | 16.7 (3.3)
Patient Health Questionnaire (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — Patient Health Questionnaire (PHQ-9) score is a standard assessment of severity of depression symptoms. (range: 0 [better], 27 [worse]). http://www.apa.org/pi/about/publications/caregivers/practice-settings/assessment/tools/patient-health.aspx
  units on a scale | 15.9 (5.2) | 16.3 (5.2) | 16.3 (5.2) | 16.2 (5.2)
CGI - Severity Score [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impression (CGI) - Severity score - standard questionnaire for severity of depression symptoms (range: 1 [less severe],7 [more severe]), https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2880930/ Population: Assessments missing for two participants at baseline.
  units on a scale
    number analyzed (Participants) | 510 | 505 | 505 | 1520
    (all) | 4.5 (1.0) | 4.6 (0.9) | 4.6 (1.0) | 4.6 (1.0)
Beck Anxiety Inventory [Mean (Standard Deviation); unit: units on a scale] — Beck Anxiety Inventory (BAI) - This is a standard questionnaire to assess anxiety of participant. The mean and standard deviation of the total score (range: 0 [low anxiety - better], 63 [higher anxiety - worse] ), https://www.beckinstitute.org/get-informed/tools-and-resources/professionals/patient-assessment-tools/ Population: Assessment missing for three participants at baseline
  units on a scale
    number analyzed (Participants) | 510 | 506 | 503 | 1519
    (all) | 18.6 (11.1) | 19.0 (11.4) | 19.7 (11.3) | 19.1 (11.3)
Arizona Sexual Experiences Scale (Female) [Mean (Standard Deviation); unit: participants] — This is a standard questionnaire for quantification of sexual dysfunction. The mean and standard deviation of the total score are presented here (range 5-30; 5 indicates better experiences, 30 indicates worse experiences) - this version is specific to females. Population: The ASEX (female) version of the questionnaire was specific to females. Not all females completed the questionnaire, therefore, the number of responders is lower than number of female participants due to missing responses.
  participants
    number analyzed (Participants) | 64 | 76 | 73 | 213
    (all) | 4.2 (1.1) | 4.2 (1.1) | 4.2 (1.2) | 4.2 (1.1)
Arizona Sexual Experiences Scale (male) [Mean (Standard Deviation); unit: participants] — This is a standard questionnaire for quantification of sexual dysfunction. Mean and standard deviation of total score are presented here (range 5-30; 5 indicates better experiences, 30 indicates worse experiences) - this version specific to males. Not all males completed the questionnaire, number of responders is lower than number of males due to missing responses. Population: The ASEX (male) version of the questionnaire was specific to males. Not all males completed the questionnaire, therefore, the number of responders is lower than number of male participants due to missing responses.
  participants
    number analyzed (Participants) | 434 | 418 | 421 | 1273
    (all) | 4.1 (1.1) | 4.1 (1.1) | 4.1 (1.2) | 4.1 (1.1)
PTSD [Count of Participants; unit: Participants] — Post-traumatic stress disorder (PTSD) determined by PTSD panel on MINI International Neuropsychiatric Interview (MINI) V6.0.0 following the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria, administered prior to randomization - current diagnosis.
  Participants | 248 | 244 | 225 | 717
EuroQol Health State Score [Mean (Standard Deviation); unit: units on a scale] — General health-related quality of life (range 0 - 100; 0 indicates worse health state, 100 indicates best possible health state) Population: Assessment missing for one participant at baseline
  units on a scale
    number analyzed (Participants) | 511 | 505 | 505 | 1521
    (all) | 54.7 (20.5) | 52.7 (19.8) | 54.0 (20.8) | 53.8 (20.4)
Quality of Life Enjoyment and Satisfaction Score [Mean (Standard Deviation); unit: units on a scale] — Quality of Life Enjoyment and Satisfaction (Q_LES_Q) Score - adjusted for percent of maximum score - measures general quality of life (percent of raw score ranges 0 - 100; 0 indicates worse quality, 100 indicates best quality)
  units on a scale | 41.4 (13.8) | 40.3 (14.8) | 40.1 (14.8) | 40.6 (14.5)
Cumulative Illness Rating Scale (CIRS) Severity Index [Mean (Standard Deviation); unit: units on a scale] — Standard questionnaire to assess comorbidities (range 0-56; 0 indicates least comorbidities [none], 56 greatest severity of comorbidities)
  units on a scale | 11.4 (5.5) | 11.1 (4.9) | 11.0 (5.1) | 11.2 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Protocol Remission of Symptoms of Major Depressive Disorder
Description: Remission of symptoms of major depression during the acute treatment phase (12 weeks) defined as a sustained clinician-rated Quick Inventory of Depressive Symptoms (QIDS-C16) of <= 5 for two consecutive visits.
Time Frame: During acute phase (12 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Switching: Bupropion-SR | Augmenting: Antidepressant + Bupropion-SR | Augmenting: Antidepressant + Aripiprazole
Number analyzed (Participants) | 511 | 506 | 505
Participants | 114 | 136 | 146
Statistical Analysis 1: Comparison: Switching: Bupropion-SR vs Augmenting: Antidepressant + Bupropion-SR; Test type: Superiority; p = 0.076, Regression, Logistic — Co-primary hypothesis: After ordering results from largest p-value to smallest (Hochberg approach) the comparison of Augmenting Antidepressant+Bupropion with Switching to Bupropion-SR was performed at the 0.05 significance level; Stratified by participating medical center; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.97 to 1.75] — Represents relative odds of remission for Augmentation Antidepressant + Bupropion-SR / Switching to Bupropion-SR
Statistical Analysis 2: Comparison: Switching: Bupropion-SR vs Augmenting: Antidepressant + Aripiprazole; Co-primary hypothesis: After ordering results form largest p-value to smallest (Hochberg approach) the comparison of Augmentation Antidepressant + Aripiprazole with Switching to Bupropion-SR was performed at the 0.025 significance level; Test type: Superiority; p = 0.018, Regression, Logistic — Co-primary hypothesis: Second ordered test after ordering largest p-value to smallest (Hochberg approach) the comparison of Augmentation Antidepressant + Aripiprazole with Switching to Bupropion-SR was performed at the 0.025 significance level; Stratified by participating medical center; Odds Ratio (OR) = 1.42, 95% CI 2-sided [1.06 to 1.89] — Represents relative odds of remission for Augmentation Antidepressant + Aripiprazole / Switching to Bupropion-SR
Statistical Analysis 3: Comparison: Augmenting: Antidepressant + Bupropion-SR vs Augmenting: Antidepressant + Aripiprazole; If either if the first two hypothesis tests for the co-primary hypotheses were significant, perform the test of Augmentation Antidepressant + Aripiprazole vs. Augmentation Antidepressant + Bupropion-SR at the 0.05 significance level; Test type: Superiority; p = 0.46, Regression, Logistic — Following the gate-keeping strategy of the analysis plan, complete the comparison of Augmentation Antidepressant + Aripiprazole vs. Augmentation Antidepressant + Bupropion-SR was evaluated at the 0.05 significance level; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.84 to 1.48] — Represents relative odds of remission for Augmentation Antidepressant + Aripiprazole / Augmentation Antidepressant + Bupropion-SR

2. Secondary Outcome: Rate of Protocol Relapse of Symptoms of Major Depression After Achieving Remission in the Acute Phase
Description: Relapse in symptoms of major depression defined as a QIDS-C16 => 11 among those achieving remission in the acute phase.
Time Frame: Within 36 weeks after randomization (initiation of treatment)
Population: The Analysis Population is the cohort of participants who met the criteria for protocol remission during the Acute Phase (first 12 Weeks of follow-up)
Measure: Count of Participants; unit: Participants
Arm/Group | Switching: Bupropion-SR | Augmenting: Antidepressant + Bupropion-SR | Augmenting: Antidepressant + Aripiprazole
Number analyzed (Participants) | 114 | 136 | 146
Participants | 26 | 35 | 37
Statistical Analysis 1: Comparison: Switching: Bupropion-SR vs Augmenting: Antidepressant + Bupropion-SR; Test type: Superiority; p = 0.70, Log Rank; Hazard Ratio (HR) = 1.36, 95% CI 2-sided [0.78 to 2.39] — Represents relative odds of relapse for Augmentation Antidepressant + Bupropion-SR / Switching to Bupropion-SR
Statistical Analysis 2: Comparison: Switching: Bupropion-SR vs Augmenting: Antidepressant + Aripiprazole; Test type: Superiority; p = 0.68, Log Rank; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.65 to 1.94] — Represents relative odds of relapse for Augmentation Antidepressant + Aripiprazole / Switching to Bupropion-SR
Statistical Analysis 3: Comparison: Augmenting: Antidepressant + Bupropion-SR vs Augmenting: Antidepressant + Aripiprazole; Test type: Superiority; p = 0.87, Log Rank; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.58 to 1.59] — Represents relative odds of relapse for Augmentation Antidepressant + Aripiprazole / Augmentation Antidepressant + Bupropion-SR

3. Secondary Outcome: Rate of Protocol Response as Reduction in Symptoms of Major Depression (>= 50% Reduction in QIDS-C)
Description: Response measured as reduction in symptom score for major depression defined as: 1. a reduction in QIDS-C16 of 50% or greater
Time Frame: During acute phase (up to 12 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Switching: Bupropion-SR | Augmenting: Antidepressant + Bupropion-SR | Augmenting: Antidepressant + Aripiprazole
Number analyzed (Participants) | 511 | 506 | 505
Participants | 319 | 332 | 375
Statistical Analysis 1: Comparison: Switching: Bupropion-SR vs Augmenting: Antidepressant + Bupropion-SR; After ordering results form largest p-value to smallest (Hochberg approach) the comparison of Augmentation Antidepressant + Bupropion with Switching to Bupropion was performed at the 0.05 significance level; Test type: Superiority; p = 0.28, Regression, Logistic; Stratified by participating medical center; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.89 to 1.50] — Represents relative odds of response for Augmentation Antidepressant + Bupropion / Switching to Bupropion
Statistical Analysis 2: Comparison: Switching: Bupropion-SR vs Augmenting: Antidepressant + Aripiprazole; After ordering results form largest p-value to smallest (Hochberg approach) the comparison of Augmentation Antidepressant + Aripiprazole with Switching to Bupropion-SR was performed at the 0.025 significance level; Test type: Superiority; p < 0.0001, Regression, Logistic; Stratified by participating medical center (site); Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.33 to 2.29] — Represents relative odds of response for Augmentation Antidepressant + Aripiprazole / Switching to Bupropion-SR
Statistical Analysis 3: Comparison: Augmenting: Antidepressant + Bupropion-SR vs Augmenting: Antidepressant + Aripiprazole; Test type: Superiority; p = 0.002, Regression, Logistic — Following the gate-keeping strategy of the analysis plan, complete the comparison of Augmentation Antidepressant + Aripiprazole with Augmentation Antidepressant + Bupropion-SR at the 0.05 significance level; Stratified by participating medical center; Odds Ratio (OR) = 1.55, 95% CI 2-sided [1.17 to 2.05] — Represents relative odds of response for Augmentation Antidepressant + Aripiprazole / Augmentation Antidepressant + Bupropion-SR

4. Secondary Outcome: Rate of Protocol Response Measured as a Change in Clinical Global Impression (CGI) - Improvement Scale
Description: Clinical assessment of a participant's level of depression and treatment response assessed by the Clinical Global Impression - Improvement (CGI -I) Scale, a 7-point clinician rating scale of improvement from baseline in severity of depression (Guy 1976). A secondary outcome measure of response was defined as achieving a score of 2 (much improved) or 1 (very much improved).
Time Frame: During acute phase (up to 12 weeks)
Population: Whole randomized cohort by intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Switching: Bupropion-SR | Augmenting: Antidepressant + Bupropion-SR | Augmenting: Antidepressant + Aripiprazole
Number analyzed (Participants) | 511 | 506 | 505
Participants | 356 | 376 | 400
Statistical Analysis 1: Comparison: Switching: Bupropion-SR vs Augmenting: Antidepressant + Bupropion-SR; Test type: Superiority; p = 0.11, Regression, Logistic — After ordering results form largest p-value to smallest (Hochberg approach) the comparison of Augmentation Antidepressant + Bupropion with Switching to Bupropion was performed at the 0.05 significance level; Stratified by participating medical center; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.95 to 1.68] — Represents relative odds of response for Augmentation Antidepressant + Bupropion / Switching to Bupropion
Statistical Analysis 2: Comparison: Switching: Bupropion-SR vs Augmenting: Antidepressant + Aripiprazole; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.001, Regression, Logistic; Stratified by participating medical center; Odds Ratio (OR) = 1.70, 95% CI 2-sided [1.26 to 2.29] — Represents relative odds of response for Augmentation Antidepressant + Aripiprazole / Switching to Bupropion-SR
Statistical Analysis 3: Comparison: Augmenting: Antidepressant + Bupropion-SR vs Augmenting: Antidepressant + Aripiprazole; Test type: Superiority; p = 0.043, Regression, Logistic — [p-value comment as in outcome 3, analysis 3]; Odds Ratio (OR) = 1.37, 95% CI 2-sided [1.01 to 1.86] — [estimate comment as in outcome 3, analysis 3]

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from the time of enrollment to withdrawal (up to 36 weeks after randomization) with one month of surveillance after withdrawal. Non-serious adverse events were collected from the time of randomization to withdrawal (up to 36 weeks after randomization).
Description: A non-serious adverse events was reported if it was among the symptoms prompted for at each scheduled follow-up or if it was a symptom assessed as possibly related to s study medication.
Groups:
- Augmenting: Antidepressant + Bupropion-SR: Augmenting: Antidepressant + Bupropion-SR
  Augmenting: Antidepressant + Bupropion-SR: Current antidepressant (either a SSRI or a SNRI or mirtazapine): Continue the dose prescribed at time of enrollment, or adjust depending on response or side effect profile for up to 36 weeks.
  And
  Bupropion-SR (Dose: 150 mg - 400 mg taken per day orally for up to 36 weeks): Initiating with bupropion-SR dose of 150 mg, then increasing dose per protocol up to 400 mg (200 mg BID), maintaining or decreasing dose for up to 36 weeks depending on response and side effect profile through the acute and continuation phases.
- Augmenting: Antidepressant + Aripiprazole: Augmenting: Antidepressant + Aripiprazole
  Augmenting: Antidepressant + Aripiprazole: Current antidepressant (either a SSRI or a SNRI or mirtazapine): Continue the dose prescribed at time of enrollment or adjust depending on response or side effect profile for up to 36 weeks.
  And
  Aripiprazole (Dose: 2 mg - 15 mg taken orally once per day for up to 36 weeks): Initiating with aripiprazole dose of 2 mg for one week, then increasing dose per protocol up to 15 mg, maintaining or decreasing dose for up to 36 weeks depending on response and side effect profile through the acute and continuation phases.
Arm/Group | Switching: Bupropion-SR | Augmenting: Antidepressant + Bupropion-SR | Augmenting: Antidepressant + Aripiprazole
All-Cause Mortality (participants affected / at risk) | 3/511 | 1/506 | 4/505
Serious Adverse Events (participants affected / at risk) | 52/511 | 57/506 | 56/505
Other Adverse Events (participants affected / at risk) | 383/511 | 369/506 | 374/505
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Switching: Bupropion-SR (N=511) | Augmenting: Antidepressant + Bupropion-SR (N=506) | Augmenting: Antidepressant + Aripiprazole (N=505)
Psychiatric disorders (total) (Psychiatric disorders) | 15 (15) | 14 (17) | 13 (16)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Alcoholism (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Drug abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Homicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Self-injurious ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Somatisation disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Substance abuse (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 8 (8) | 10 (11) | 5 (5)
Suicide attempt (Psychiatric disorders) | 3 (3) | 1 (1) | 3 (3)
Nervous system disorders (total) (Nervous system disorders) | 7 (7) | 3 (4) | 3 (4)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Drug withdrawal headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 2 (3) | 0 (0)
Serotonin syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders (total) (Gastrointestinal disorders) | 3 (3) | 2 (3) | 2 (2)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperaldosteronism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions (total) (General disorders) | 4 (6) | 2 (2) | 5 (6)
Adverse drug reaction (General disorders) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 3 (4)
Device malfunction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hernia obstructive (General disorders) | 1 (3) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders (total) (Cardiac disorders) | 7 (7) | 4 (4) | 8 (8)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Nodal rhythm (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Bladder perforation (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Accident at work (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (3)
Infections and infestations (total) (Infections and infestations) | 6 (6) | 10 (11) | 12 (14)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis of male external genital organ (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eczema infected (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infectious colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infective tenosynovitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 4 (4) | 3 (3)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Alcohol detoxification (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Drug detoxification (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Switching: Bupropion-SR (N=511) | Augmenting: Antidepressant + Bupropion-SR (N=506) | Augmenting: Antidepressant + Aripiprazole (N=505)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders (Cardiac disorders) | 4 (4) | 2 (2) | 3 (3)
Congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0/0 (0)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 4 (4) | 11 (12) | 1 (1)
Eye disorders (Eye disorders) | 5 (5) | 10 (10) | 12 (14)
Gastrointestinal disorders (Gastrointestinal disorders) | 189 (305) | 157 (288) | 147 (230)
General disorders and administration site conditions (General disorders) | 82 (100) | 73 (97) | 105 (115)
Hepatobiliary disorders (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations (Infections and infestations) | 20 (21) | 10 (13) | 11 (12)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (2) | 11 (12) | 9 (10)
Investigations (Investigations) | 25 (28) | 38 (41) | 72 (81)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 114 (134) | 95 (111) | 113 (142)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 20 (21) | 10 (10) | 17 (20)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Nervous system disorders (Nervous system disorders) | 218 (383) | 235 (426) | 239 (433)
Psychiatric disorders (Psychiatric disorders) | 224 (393) | 200 (349) | 176/176 (270)
Renal and urinary disorders (Renal and urinary disorders) | 8 (8) | 9 (10) | 6 (6)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (2) | 9 (9) | 7 (7)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 5 (5) | 10 (12)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 50 (63) | 48 (58) | 38 (45)
Social circumstances (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
Vascular disorders (Vascular disorders) | 7 (8) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes